CLINICAL TRIAL: NCT04506346
Title: Risk Prediction of Difficult Tracheal Intubation in Obstructive Sleep Apnea Hypopnea Syndrome Patient (OSAHS) Undergoing Uvulo-palato-pharyngoplasty
Brief Title: Risk Prediction of Difficult Tracheal Intubation in OSAHS Patient
Acronym: OSAHS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XMLX201824
Record Dates: First submitted 2020-02-01; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Difficult Intubation; Airway Obstruction
Keywords: airway management; obstructive sleep apnea hypopnea syndrome; risk predictive model
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OSAHS: patients with OSAHS, undergoing UPPP
  Interventions: Diagnostic Test: difficult tracheal intubation

INTERVENTIONS:
Diagnostic Test: difficult tracheal intubation — Grade Ⅲ or Ⅳ according to Cormach-Lehane Grading of laryngoscopic view

SUMMARY:
This study evaluates the risk factors for difficult tracheal intubation in in obstructive sleep apnea hypopnea syndrome(OSAHS) patients undergoing uvulo-palato-pharyngoplast(UPPP)

DETAILED DESCRIPTION:
OSAHS patients are high risk group of difficult tracheal intubation. In clinical application, unexpected difficult tracheal intubation is not rare. Difficult airway is a significant problem to these patients and the physicans in terms of mortality and morbidity.

This study collects risk factors as physical examinations（including modified Mallampati grade, neck circumference, lateral clinical craniofacial assessment and body mass index ,BMI）, Stopbang scores, polysommographic parameters (including apnea-hypopnea index, AHI and lowest SpO2, LSpO2), and special radiographic parameters in head and neck region. By using statistics method, predictive model to manage risks would be established.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as OSAHS.
* receive UPPP under general anesthesia in Beijing Tsinghua Changgung Hospital
* ASA grade I or II

Exclusion Criteria:

* ASA grade III or above
* had received UPPP
* had fore-teeth loosed
* obstructive sleep apnea hypopnea were caused by hypothyroidism, acromegaly, or vocal cord paralysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate or severe obstructive sleep apnea hypopnea syndrome, which means apnea-hypopnea index( AHI) >15/h and lowest SpO2(LSpO2)<85% in polysommographic test.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Difficult Tracheal Intubation | 1min After tracheal intubation
  Grade Ⅲ or Ⅳ according to Cormach-Lehane Grading of laryngoscopic view

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhang, MD, Study Chair — department of anesthesia
Locations (1):
- YAN SIYI, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No